CLINICAL TRIAL: NCT06692959
Title: A Phase II Trial of Neoadjuvant PD-1 Vaccine PD1-Vaxx in Operable MSI High Colorectal Cancer
Acronym: Neo-POLEM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Australasian Gastro-Intestinal Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79361
Record Dates: First submitted 2024-11-07; First posted 2024-11-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: PD-1 Vaccine; Operable Colorectal Cancer; Neo-adjuvant
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a phase II, Bayesian Optimal Design, single arm, one cohort, open label, multi-centre study of neoadjuvant PD-1 vaccine PD1-Vaxx and surgical resection in adult patients with operable MSI-high colorectal cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD1-Vaxx (Experimental): All patients will be administered PD1-Vaxx intramuscularly into the deltoid region of the upper arm on days 1,15 and 29. Patients will undergo resection surgery within 21 days, but up to 42 days of completing trial treatment.
  Interventions: Drug: PD-1 vaccine IMU-201 (PD1-Vaxx)

INTERVENTIONS:
Drug: PD-1 vaccine IMU-201 (PD1-Vaxx) — Investigational Medicinal Product (IMP) PD1-Vaxx is supplied as lyophilized drug substance APi2568, which is a B-cell epitope (amino acids 92-110 from PD-1) linked to a promiscuous T-cell epitope (amino acid residues 288-302 from measles virus fusion protein) via a 4-amino acid linker (G-P-S-L). IMU-201 is combined with water for Injection (WFI) and is emulsified with Montanide ISA 51 VG adjuvant to produce PD1-Vaxx.

SUMMARY:
The aim of Neo-POLEM is to determine the rate of Major Pathological Response (MPR) of <10% viable tumour cells after administering neoadjuvant PD-1 vaccine IMU-201 (PD1-Vaxx), as measured by percentage change pre- and post-treatment in operable MSI high CRC patients.

All patients will be administered three doses of the PD1-Vaxx prior to resection surgery and will be followed up for a minimum of 2 years.

DETAILED DESCRIPTION:
This is a phase II, Bayesian Optimal Design, single arm, one cohort, open label, multi-centre study of neoadjuvant PD-1 vaccine PD1-Vaxx and surgical resection in adult patients with operable MSI-high colorectal cancer. All patients will be administered PD1-Vaxx intramuscularly into the deltoid region of the upper arm on days 1,15 and 29. Patients will undergo resection surgery within 21 days, but up to 42 days of completing trial treatment. The resection sample will be examined locally for pathological response within 28 days of surgical resection. Patient will then remain in active follow up for up to 2 years. Once the last patient has completed their last visit a check will be made on all patients to confirm their recurrence and survival status.

The aim of the trial is to determine the major pathological response rates after administering neoadjuvant PD-1 vaccine PD1-Vaxx in operable MSI-high CRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed and dated a written informed consent form. This must be performed before the performance of any protocol related procedures that are not part of the normal care.
2. Patients must be willing and able to comply with the schedule visits, treatment schedules, laboratory tests and other requirements of the study.

   Target Population
3. Histologically confirmed adenocarcinoma cancer of the colon and high rectum.
4. ECOG Performance status 0 or 1
5. Measurable disease per RECIST 1.1 criteria
6. Tumour tissue from a colonoscopy must be provided for biomarker analysis. Archival tumour tissue is mandatory for biomarker analysis. If no sample is available, patients will have the option to agree to acquisition of additional tumour tissue during the screening period for future biomarker analyses...
7. In order in to be entered into the study, patients must be classified as MSI-High (confirmation of MMR deficiency or MSI-H).
8. Stage II (T3-T4 N0) III (any T, N1 or N2, M0) Colorectal cancer
9. Radiological evidence of operable CRC, determined by local MDT, usually CT scan.
10. Treatment naive patients (no prior anti CRC therapy).
11. Screening laboratory values must meet the following criteria

    1. Neutrophils ≥ 1.5x 109/L
    2. Platelets ≥ 100 x 109/L
    3. Haemoglobin ≥ 9.0 g/dl
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance 'CrCl' > 50 mL/min (using the Cockcroft Gault formula):

       * Female CrCl = (140 - age in years) x weight (kg) x 1.04 serum creatinine (µmol/l)
       * Male CrCl = (140 - age in years) x weight (kg) x 1.23 serum creatinine in µmol
    5. Total bilirubin ≤ 1.5 x ULN; for patients with documented/suspected Gilbert's disease, bilirubin ≤3 x ULN
    6. AST ≤1.5 x ULN
    7. ALT ≤1.5 x ULN

    Age and Reproductive Status
12. Age ≥ 18 years
13. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study drug.
14. Women must not be breastfeeding.
15. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception, as indicated in the informed consent form. Contraception must be used for the duration of treatment and for a period of 180 days after last dose of study drug.
16. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception, as indicated in the informed consent form for a period of 180 days. Men who are sexually active with WOCBP must continue contraception for 180 days after the last dose of investigational drug (combination or monotherapy). In addition, male patients must be willing to refrain from sperm donation during this time.
17. Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, and still must undergo pregnancy testing as described in this section.

    Exclusion Criteria:
18. History of severe allergic reactions (i.e., Grade 4 allergy, anaphylactic reaction from which the patient did not recover within 6 hours of institution of supportive care) to any unknown allergens or any components of the PD-1 vaccine formulations.
19. Distant metastases or peritoneal nodules (M1)
20. Active or prior documented autoimmune disease (including inflammatory bowel disease, coeliac disease, and Wegener syndrome).
21. Any concurrent chemotherapy or biologic or hormonal therapy for CRC treatment. Concurrent use of hormones for non-cancer- related conditions (e.g. insulin for diabetes and hormone replacement therapy) is acceptable.
22. History of primary immunodeficiency, solid organ transplantation, or previous clinical diagnosis of tuberculosis.
23. If they are positive for hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
24. If they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
25. Receipt of live, attenuated vaccine within 28 days prior to the first dose of PD-1 vaccine PD1-Vaxx (patients, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of Investigational Medicinal Product (IMP)).
26. Other invasive malignancy within two years except for non-invasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured. Cancer patients with incidental histological findings of prostate cancer (tumour/node/metastasis stage of T1a or T1b or prostate-specific antigen ˂10) who have not received hormonal treatment may be included.
27. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement or compromise the ability of the patient to give written informed consent.
28. Any condition that, in the opinion of the investigator or sponsor, would interfere with the evaluation of the investigational product or interpretation of patient safety or study results.
29. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisolone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisolone equivalents are permitted in the absence of active autoimmune disease.
30. Systemic antibiotic treatment within 7 days prior to the start of trial treatment.
31. Patients with a documented history of pneumonitis, regardless of the cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) rates after administering neoadjuvant PD-1 vaccine | At surgery
  Proportion of participants with MPR (determined by ≤10% viable tumour cells after receiving PD1-Vaxx).

SECONDARY OUTCOMES:
Safety of PD-1 vaccine PD1-Vaxx in the neo-adjuvant setting | From first vaccine dose until 100 days after the last study treatment
  Adverse events graded according to CTCAE v5
Rate of complete response after receiving PD1-Vaxx | At surgery
  Proportion of participants with complete response (no viable tumour cells after receiving PD1-Vaxx).
Objective response rate | 21 days after last vaccine
  Overall Response Rate (ORR) by RECIST 1.1
Disease free survival | From surgery until completion of 2 year follow up
  Disease-free survival
Overall survival | From enrolment to completion of 2 years follow up
  Overall survival
Claviend-Dindo | 30 days post surgery
  Clavien-Dindo grading
Health-related quality of life | 21 days after last vaccine
  EORTC QLQ-C30
Health-related quality of life | 21 days after last vaccine
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - The Christie NHS Foundation Trust, Manchester